CLINICAL TRIAL: NCT03577301
Title: Comparative Effectiveness Trial of Clinic-Based Delivery of an HIV Risk Reduction Intervention for Young Men Who Have Sex With Men (YMSM)
Brief Title: Young Men's Health Project Targeting HIV Risk Reduction and Substance Abuse
Acronym: YMHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Sylvie Naar, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ATN145
Record Dates: First submitted 2018-04-06; First posted 2018-07-05 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
Keywords: HIV; Intervention; Men Who Have Sex with Men (MSM); PrEP; YMHP; YMSM
MeSH Terms: conditions — HIV Infections; Homosexuality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clinic-based Delivery (Active Comparator): Participants will receive the intervention in person following HIV counseling and testing. The intervention involves completion of the 4 YMHP sessions and the delivery of pre-exposure prophylaxis (PrEP) information and navigation services to interested participants. This arm is closed to enrollment.
  Interventions: Behavioral: Clinic-based Delivery
- Remote Delivery (Active Comparator): Participants will receive the intervention by remote delivery following HIV counseling and testing. Just as the clinic-based participants, he intervention involves completion of the 4 YMHP sessions and the delivery of pre-exposure prophylaxis (PrEP) information and navigation services to interested participants. This arm is closed to enrollment.
  Interventions: Behavioral: Remote Delivery
- Multi-modal Delivery (Active Comparator): A 4 session MI intervention. Session 1 is always delivered in person immediately after baseline. Session 2-4 can be delivered in person or remotely based upon youth preference. This arm is open to enrollment as of 11/15/2019.
  Interventions: Behavioral: Multi-modal Delivery
- Treatment as Usual (No Intervention): Treatment as usual control = individual HIV testing with referrals and link age to care as provided by the sites under routine circumstances. This arm is open to enrollment as of 11/15/2019.

INTERVENTIONS:
Behavioral: Clinic-based Delivery — A minimum of 2 community health workers (CHWs) will be trained to deliver clinic-based intervention sessions.
  Arms: Clinic-based Delivery
Behavioral: Remote Delivery — A minimum of 2 community health workers (CHWs) will be trained to deliver intervention sessions to the participant in a location remote from the clinic setting.
  Arms: Remote Delivery
Behavioral: Multi-modal Delivery — A minimum of 2 community health workers (CHWs) will be trained to deliver clinic-based or remote intervention sessions. First MI session is in person immediately after baseline. Sessions 2-4 can be delivered in person or remotely based on youth preference.
  Arms: Multi-modal Delivery

SUMMARY:
YMHP is a counseling intervention program for which the goals are to better understand HIV-prevention focused self-management behaviors among HIV-negative YMSM, and to study the implementation of YMHP to improve portability and scalability. The clinic sites will help investigators to assess and address practical problems at the frontline of service provision to pave the way for a comprehensive program to reduce HIV infection among YMSM that reflects the complexities of real world adolescent HIV clinics.

DETAILED DESCRIPTION:
1. Adapt YMHP for clinic and phone delivery by existing HIV clinic staff community health workers (CHWs), who work with YMSM ages 15-24. Investigators will conduct focus groups with staff to obtain input on how best to implement YMHP to maximize feasibility, acceptability, and sustainability, as well as issues with adapting the YMHP for delivery to YMSM ages 15-18 and for phone delivery.
2. Compare the effectiveness of clinic-based versus phone-based delivery of YMHP in the context of health care access. In order to inform future implementation, investigators will test the effectiveness of YMHP delivered via these two modalities.

   1. Assess the cost-effectiveness of both delivery formats of YMHP to enhance the likelihood of uptake of this best evidence intervention. The hypothesis is that phone-based will be more cost-effective than clinic-based
   2. Assess the Five Components of the Self-Management Model and how these components vary over time, are directly improved by the interventions, and mediate intervention effects.
3. Test a sustainable model of YMHP implementation in real world adolescent clinics. Investigators will utilize local supervisors within the clinic setting to sustain the CHWs fidelity to delivering the motivational interviewing (MI)-based YMHP intervention. Fidelity will be monitored throughout the trial and assessments and qualitative interviews will be conducted with key stakeholders to determine the barriers and facilitators of YMHP implementation utilizing the Exploration, Preparation, Implementation, Sustainment model (EPIS).

Aims will be achieved over two phases of the study.

Phase I: Investigators will conduct research (Exploration and Preparation phases of EPIS model) to obtain implementation feedback to best adapt YMHP for clinic-based CHWs, further incorporate PrEP navigation services, and expand the YMHP protocol to be relevant for Telephone-based Motivational Interviewing (TBMI). We will train a minimum of 2 CHWs at each clinic drawing on the Implementation Science Core (ISC) to apply best-practices in training. Once CHWs demonstrate competence according to the Motivational Interviewing Treatment Integrity (MITI), Phase 2 will begin.

Phase II: Personnel will recruit and enroll 180 YMSM, ages 15-24, 60 at each of the three sites. Sessions will be audio-recorded for MITI fidelity coding, and CHWs and supervisors will be given implementation support throughout. Prior to implementation, immediately at the conclusion of the intervention delivery phase, and one year after, the ISC will conduct interviews with CHWs, supervisors, and clinic leaders to obtain information about the barriers and facilitators of implementation and sustainment.

Target n: 180 YMSM across three sites (60 per site).

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative test result from the past 90 days
* 15-24 years of age
* Born biologically male or currently identifying as male
* Sex with men in the past 90 days
* ≥ 3 days of illicit drug use in the past 90 days
* ≥ 1 episode of Condomless Anal Sex (CAS) in the past 90 days, or a positive STI test result in the past 90 days.
* Able to communicate in English

Exclusion Criteria:

* Serious cognitive or psychiatric impairments
* Currently taking Truvada as Pre-Exposure Prophylaxis (PrEP)

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Born biologically male or currently identifying as male
Enrollment: 83 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naar, PhD, Principal Investigator — Florida State University
Locations (3):
- United States (3):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Wayne State University, Detroit, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinic-based Delivery | Remote Delivery | Multi-modal Delivery | Treatment as Usual
Started | 24 | 21 | 16 | 22
Completed | 24 | 21 | 16 | 22
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinic-based Delivery | Remote Delivery | Multi-modal Delivery | Treatment as Usual | Total
Number analyzed (Participants) | 24 | 21 | 16 | 22 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 7 | 3 | 1 | 12
  Between 18 and 65 years | 23 | 14 | 13 | 21 | 71
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 24 | 21 | 16 | 22 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 7 | 9 | 6 | 9 | 31
  Race/Ethnicity: Latino | 9 | 6 | 8 | 7 | 30
  Race/Ethnicity: White | 4 | 3 | 2 | 5 | 14
  Race/Ethnicity: Other/Multiracial | 4 | 3 | 0 | 1 | 8
Sexual Identity [Count of Participants; unit: Participants]
  Gay/Queer | 18 | 17 | 12 | 17 | 64
  Bisexual/Other | 6 | 4 | 4 | 5 | 19
Site [Count of Participants; unit: Participants]
  Site 1 | 4 | 5 | 2 | 5 | 16
  Site 2 | 12 | 11 | 14 | 13 | 50
  Site 3 | 8 | 5 | 0 | 4 | 17
Relationship Status [Count of Participants; unit: Participants]
  Single | 16 | 14 | 6 | 11 | 47
  Partnered | 8 | 7 | 10 | 11 | 36
Education [Count of Participants; unit: Participants]
  4-Year College Degree or more | 6 | 2 | 2 | 5 | 15
  Some college of Associates Degree | 10 | 10 | 12 | 13 | 45
  Some High School | 8 | 9 | 2 | 4 | 23

OUTCOME MEASURES:

1. Primary Outcome: Illicit Drug Use Days
Description: The self-reported number of illicit drug use days (not including marijuana) in the past 30 days
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Clinic-based Delivery | Remote Delivery | Multi-modal Delivery | Treatment as Usual
Number analyzed (Participants) | 24 | 21 | 16 | 22
Number of Days
  Use at Baseline | 3.17 (4.10) | 3.10 (7.37) | 3.25 (5.99) | 2.86 (6.76)
  Use at 3 Months | 9.00 (19.16) | 5.12 (10.89) | 2.55 (5.66) | 9.21 (29.62)
  Use at 6 Months | 9.64 (24.38) | 5.93 (16.04) | 3.23 (9.03) | 2.64 (6.17)
  Use at 9 Months | 1.58 (3.70) | 3.46 (8.35) | 7.45 (23.09) | 10.93 (34.99)
  Use at 12 Months | 9.91 (27.70) | 3.80 (9.27) | 1.00 (1.89) | 1.33 (1.21)
Statistical Analysis 1: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.35, Negative Binomial Regression; Model testing whether condition predicted illicit drug use at 3 months; Wald Chi Square = 3.30
Statistical Analysis 2: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.58, Negative Binomial Regression; Model testing whether condition predicted illicit drug use at 6 months; Wald Chi Square = 1.97
Statistical Analysis 3: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.64, Negative Binomial Regression; Model testing whether condition predicted illicit drug use at 9 months; Wald Chi Square = 1.68
Statistical Analysis 4: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.76, Negative Binomial Regression; Model testing whether condition predicted illicit drug use at 12 months; Wald Chi Square = 1.15

2. Primary Outcome: Condomless Anal Sex Acts
Description: The self-reported number of condomless anal sex acts with male partners in the last 30 days prior to assessment point.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Acts in the past 30 days
Arm/Group | Clinic-based Delivery | Remote Delivery | Multi-modal Delivery | Treatment as Usual
Number analyzed (Participants) | 24 | 21 | 16 | 22
Acts in the past 30 days
  Baseline | 5.9 (4.91) | 4.5 (8.6) | 6.9 (8.98) | 10.0 (14.54)
  3 Month | 3.1 (4.44) | 5.9 (12.81) | 6.8 (10.20) | 10.2 (20.20)
  6 Month | 5.4 (8.18) | 4.4 (10.57) | 8.9 (13.74) | 10.6 (23.93)
  9 Month | 11.0 (14.75) | 13.6 (30.07) | 13.2 (18.19) | 20.6 (48.34)
  12 Month | 10.8 (18.30) | 2.3 (5.58) | 11.9 (16.98) | 1.2 (1.30)
Statistical Analysis 1: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.38, Negative Binomial Regression; Model testing whether condition predicted condomless anal sex acts at 3 months; Wald Chi Square = 3.08
Statistical Analysis 2: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.74, Negative Binomial Regression; Model testing whether condition predicted condomless anal sex acts at 6 months; Wald Chi Square = 1.26
Statistical Analysis 3: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.74, Negative Binomial Regression; Model testing whether condition predicted condomless anal sex acts at 9 months; Wald Chi Square = 1.27
Statistical Analysis 4: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.300, Negative Binomial Regression; Model testing whether condition predicted condomless anal sex acts at 12 months; Slope = 3.66

3. Primary Outcome: Marijuana Use Days
Description: The self-reported number of marijuana use days in the past 30 days prior to assessment point.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Clinic-based Delivery | Remote Delivery | Multi-modal Delivery | Treatment as Usual
Number analyzed (Participants) | 24 | 21 | 16 | 22
Number of Days
  Baseline | 31.38 (34.01) | 34.09 (38.48) | 32.00 (35.40) | 19.00 (29.30)
  3 Month | 40.00 (37.21) | 32.75 (36.56) | 26.00 (32.66) | 20.16 (28.71)
  6 Month | 41.71 (38.43) | 32.57 (35.67) | 28.77 (32.72) | 19.50 (28.25)
  9 Month | 42.00 (41.60) | 33.08 (35.44) | 22.27 (30.05) | 24.71 (34.73)
  12 Month | 41.82 (36.61) | 37.20 (38.60) | 34.80 (38.01) | 18.50 (24.07)
Statistical Analysis 1: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.73, Negative Binomial Regression; Model testing whether condition predicted marijuana use days at 3 months; Wald Chi Square = 1.30
Statistical Analysis 2: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.64, Negative Binomial Regression; Model testing whether condition predicted marijuana use days at 6 months; Wald Chi Square = 1.68
Statistical Analysis 3: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.89, Negative Binomial Regression; Model testing whether condition predicted marijuana use days at 9 months; Wald Chi Square = 0.64
Statistical Analysis 4: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.78, Negative Binomial Regression; Model testing whether condition predicted marijuana use days at 12 months; Wald Chi Square = 1.08

4. Secondary Outcome: Alcohol Use Days
Description: The self-reported number of alcohol use days in the past 30 days
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Clinic-based Delivery | Remote Delivery | Multi-modal Delivery | Treatment as Usual
Number analyzed (Participants) | 24 | 21 | 16 | 22
Number of Days
  Baseline | 20.17 (17.82) | 13.71 (15.35) | 17.62 (20.03) | 17.27 (15.22)
  3 Month | 20.60 (17.52) | 12.06 (12.54) | 13.45 (13.57) | 16.89 (15.49)
  6 Month | 18.78 (18.63) | 9.78 (10.49) | 10.15 (11.01) | 17.36 (15.96)
  9 Month | 15.00 (14.34) | 14.61 (15.84) | 13.27 (17.27) | 17.43 (14.05)
  12 Month | 20.91 (23.34) | 13.50 (22.15) | 22.33 (18.49) | 15.30 (23.76)
Statistical Analysis 1: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.50, Negative Binomial Regression; Model testing whether condition predicted alcohol use days at 3 months; Wald Chi Square = 2.37
Statistical Analysis 2: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.34, Negative Binomial Regression; Model testing whether condition predicted alcohol use days at 6 months; Wald Chi Square = 2.98
Statistical Analysis 3: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.66, Negative Binomial Regression; Model testing whether condition predicted alcohol use days at 9 months; Wald Chi Square = 1.59
Statistical Analysis 4: Comparison: Clinic-based Delivery vs Remote Delivery vs Multi-modal Delivery vs Treatment as Usual; Test type: Superiority; p = 0.43, Negative Binomial Regression; Model testing whether condition predicted alcohol use days at 12 months; Wald Chi Square = 2.74

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Clinic-based Delivery | Remote Delivery | Multi-modal Delivery | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21 | 0/16 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/16 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/16 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03577301/Prot_001.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT03577301/SAP_002.pdf
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT03577301/ICF_003.pdf